CLINICAL TRIAL: NCT05062057
Title: Menopause Racing Heart Study
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor of Pharmacy Practice, Indiana University
Other Study IDs: 12409
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Menopause Related Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Estradiol; estrone; thyroid-stimulating hormone; C-reactive protein; interleukin-6; leptin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Palpitations: n=15 peri- and postmenopausal women with self-reported palpitations within 2 weeks prior to enrollment
  Interventions: Device: Adhesive ambulatory ECG recording patches
- No palpitations: n=15 peri- and postmenopausal women with no self-reported palpitations within 6 months prior to enrollment
  Interventions: Device: Adhesive ambulatory ECG recording patches

INTERVENTIONS:
Device: Adhesive ambulatory ECG recording patches — All women in both groups will undergo sequential placement of two 14-day adhesive ambulatory ECG recording patches for a total of 28 days of ECG recording

SUMMARY:
Palpitations occur in more than 25% of women as they approach menopause and after menopause. However, the etiology of menopausal palpitations has not been studied, and it is unknown whether palpitations in menopausal women are caused by underlying arrhythmias or other electrocardiographic (ECG) abnormalities.

Objective:

1. The primary objective of this exploratory pilot study is to assess whether arrhythmias and/or other ECG abnormalities underlie symptomatic palpitations in peri- and postmenopausal women 2 The secondary objective is to better understand women's palpitations symptom experiences (describe the symptom, its dimensions (frequency, severity, distress, duration, temporal pattern, aggravating/alleviating factors), and any attempted or actual healthcare utilization related to the symptom (provider contacts, discussions, referrals; laboratory or other tests).

In this study, 30 peri- and post-menopausal women will be enrolled to determine if they have underlying arrhythmias or other ECG abnormalities. n=15 peri/postmenopausal women who describe palpitations within the previous 2 weeks and a control group of n=15 peri/postmenopausal women who have not experienced palpitations within 6 months will be enrolled. All participants will undergo placement of a 14-day adhesive ECG monitoring patch [(Carnation Ambulatory Monitoring (CAM) patch, Bardy Diagnostics] on their chest. After wearing the patch for 14 days, the patch will be removed, and a 2nd 14-day patch will be placed, for a total of 28 days of ECG recording. Data from the adhesive ECG patches will be uploaded and an assessment of arrhythmias and other ECG changes will be made. In addition, all participants will undergo a semi-structured interview to obtain information on their palpitations symptoms experience.

Changes in study procedure:

1. To reduce participant and staff burden and costs, in April 2023, we reduced the ECG wear time to 14 days and eliminated study visit 3. We did this because the ECH patches did not always adhere well to the skin, necessitating extra study visits, extra patches, and additional costs.
2. Because of the COVID-19 pandemic delays in study initiation and the ECG issues, we recruited 15 rather than the originally planned 20 women in each group. The new sample size was consistent with our limited funding, limited staff resources, and the pilot nature of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 40-62 years
2. Upper limit of 62 years because this is 10 years past the median age at menopause, which is the age range when most women experience menopause symptoms
3. Peri-menopausal women

   * Defined as no menses in the past 3 months or menses in the past 3 months but cycles are less regular (as self-reported by the women)20
4. Postmenopausal women

   * No menses for 12 months or longer
5. Women with surgical menopause will be included
6. Willing to wear the adhesive heart monitor on their chest for 28 days
7. Palpitations group: women who have reported palpitations within the previous 2 weeks
8. Control group: Women who report having no palpitations within the past 6 months
9. Completion of 2-week symptom diary

Exclusion Criteria:

1. Pregnant
2. Breastfeeding
3. History of arrhythmias (with the exception of sinus bradycardia, sinus arrhythmia or sinus tachycardia)
4. History of stroke
5. History of heart failure
6. Permanent pacemaker
7. Taking antiarrhythmic drugs (with the exception of ß-blockers, diltiazem or verapamil)
8. Known skin allergies (CAM patches are contraindicated)
9. Family history of skin allergies (CAM patches are contraindicated)

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Peri- and postmenopausal women between the ages of 40 and 62 years who: 1) Self-report palpitations within the previous 2 weeks prior to enrollment (Palpitations group) and 2) Have no self-reported palpitations within 6 months prior to enrollment (Control group)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Arrhythmias | 28 days
  Incidence and nature of arrhythmias in peri- and postmenopausal women who report symptomatic palpitations. Arrhythmias to be assessed include, but are not limited to:
  * Accelerated idioventricular rhythm
  * AF
  * Atrial flutter
  * Atrial tachycardia
  * Atrioventricular blocks (2nd and 3rd degree)
  * Junctional rhythm
  * Junctional tachycardia
  * Premature atrial complexes (PACs)
  * PVCs, including couplets, bigeminy, trigeminy
  * Sinus tachycardia
  * Supraventricular tachycardia (AV nodal reentrant tachycardia, AV reentrant tachycardia)
  * Ventricular tachycardia (monomorphic and polymorphic)
  * Any other abnormal rhythms discovered

SECONDARY OUTCOMES:
Moment-to-moment self-report of palpitations events recorded through an event marker button | 28 days
Narrative descriptions of women's symptom experiences | 28 days
  Symptom dimensions (e.g., frequency, severity, temporal pattern) and treatment-seeking (e.g., reports to healthcare professionals, tests, ER visits)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (1):
- Indiana CTSI Clinical Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified subject data will be shared with other investigators upon request